CLINICAL TRIAL: NCT02526602
Title: Preservation of Endopelvic Fascia During Radical Prostatectomy: Effects on Postoperative Incontinence and Impotence. Randomized Clinical Trial.
Brief Title: Preservation of Endopelvic Fascia: Effects on Postoperative Incontinence and Impotence. Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R15043
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Prostatic Neoplasms; Urinary Incontinence; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence; Erectile Dysfunction | interventions — Preservation, Biological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preservation (endopelvic fascia) (Experimental): During robotic assisted laparoscopic radical prostatectomy endopelvic fascia are preserved.
  Interventions: Procedure: Preservation (endopelvic fascia)
- Opening (endopelvic fascia) (Active Comparator): During robotic assisted laparoscopic radical prostatectomy endopelvic fascia are opened.
  Interventions: Procedure: Opening (endopelvic fascia)

INTERVENTIONS:
Procedure: Preservation (endopelvic fascia) — Robotic assisted radical prostatectomy with preserving of endopelvic fascia
  Arms: Preservation (endopelvic fascia)
Procedure: Opening (endopelvic fascia) — Robotic assisted radical prostatectomy with opening of endopelvic fascia
  Arms: Opening (endopelvic fascia)

SUMMARY:
Urinary incontinence and impotence are typical disturbances after radical prostatectomy. Although, several surgical methods are developed to decrease these disturbances, 8% and 50% of the patients suffer from permanent urinary incontinence and impotence, respectively.

Previously two studies have shown that endopelvic fascia preservation may decrease postoperative incontinence and impotence rates. Unfortunately these studies are retrospective decreasing their reliability.

The present study is prospective and randomized clinical trial. The investigators are going to randomize 180 patient to preservation and opening the endopelvic fascia groups. Functional and oncological results are followed up to 1 year after surgery.

DETAILED DESCRIPTION:
180 patients going to radical prostatectomy as treatment of prostate cancer will be randomized 1:1 to two study arms: In the other arm endopelvic fascia are preserved during the operation, in the other arm the fascia are opened.

After the operation urinary continence and erection function are compared between the study arms. Additionally the investigators will study oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Localized prostate cancer
* Planned nerve-sparing robotic radical prostatectomy
* Gleason score 7 or less

Exclusion Criteria:

* Previous prostate surgery (TURP, TUIP, laser...)
* Planned lymphadenectomy
* T3 cancer

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence | 1 year
  EPIC-26 questionnaire preoperatively and 3 and 12 months after surgery
Erectile function | 1 year
  EPIC-26 questionnaire preoperatively and 3 and 12 months after surgery

SECONDARY OUTCOMES:
Complications | 1 year
  Clavien-Dindo classification
Oncologic results: positive surgical margin rate | 1 year
  Positive surgical margin rate as reported in pathological analysis of the removed prostate

CONTACTS AND LOCATIONS:
Overall Officials: Jarno Riikonen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siltari A, Riikonen J, Murtola TJ. Preservation of Endopelvic Fascia: Effects on Postoperative Incontinence and Sexual Function - A Randomized Clinical Trial. J Sex Med. 2021 Feb;18(2):327-338. doi: 10.1016/j.jsxm.2020.11.003. Epub 2020 Dec 23. PMID 33358241